CLINICAL TRIAL: NCT06969417
Title: Comparative Efficacy of Pregabalin and Lacosamide in Patients With Herpes Zoster and Post Herpetic Neuralgia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CMH Kharian Medical College (Other Government)
Responsible Party: Principal Investigator, Mushayada Irshad, Dr Mushayada Irshad, CMH Kharian Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CKMC/IERB/AC-00225
Record Dates: First submitted 2025-05-05; First posted 2025-05-13 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Herpes Zoster (HZ); Post Herpetic Neuralgia (PHN)
MeSH Terms: conditions — Herpes Zoster; Neuralgia, Postherpetic | interventions — Pregabalin; Lacosamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Active Comparator): Group A will receive Cap Pregabalin, the first intervention
  Interventions: Drug: Pregabalin
- Group B (Experimental): Group B will receive Tab Lacosamide
  Interventions: Drug: Lacosamide

INTERVENTIONS:
Drug: Pregabalin — o Group A will receive Cap Pregabalin 150mg oral OD for 4 weeks
  Arms: Group A
Drug: Lacosamide — o Group B will receive Tab Lacosamide 100mg oral BD for 4 weeks
  Arms: Group B

SUMMARY:
Post-herpetic neuralgia (PHN) is the most significant complication of herpes zoster caused by reactivation of latent Varicella-Zoster virus (VZV). PHN is characterized by neuropathic pain lasting beyond the resolution of the rashes. Post herpetic neuralgia (PHN) represents a potentially debilitating and often undertreated form of neuropathic pain that disproportionately affects vulnerable populations, including the elderly and the immunocompromised. PHN pain is typically localized, unilateral and chronic, but may be constant, intermittent, spontaneous and/or evoked. PHN is likely to interfere with sleep and daily activities.

Pregabalin is a gabapentinoid licenced for treatment of neurological disorders. It is one of the earlier drugs approved by the US Food and Drug Administration (2004) for the treatment of painful diabetic neuropathy and postherpetic neuralgia (PHN). Lacosamide (LCM) was approved in 2008 in the European Union and in the United States as adjunctive therapy for the treatment of focal-onset seizures with or without secondary generalization in adults and adolescents with epilepsy. Its efficacy has also been proven in neuropathic pain.

Although Pregabalin and Lacosamide have proven effective in various neuropathic pain disorder, comparative studies specifically for PHN remain scarce. This study aims to compare the efficacy of Pregabalin and Lacosamide in PHN patients, addressing the current gap in literature and providing clinically relevant insights to optimize treatment selection.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed cases of herpes zoster suffering from postherpetic neuralgia
* Ages: 18 to 50
* Both male and female

Exclusion Criteria:

* Lack of consent
* Patient already taking pain killers for post herpetic neuralgia
* Patients suffering from other systemic illness

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | 4 weeks
  Pain intensity will be measured before and after treatment with help of Visual Analog Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Usman Nawaz, MBBS, Mphil, PhD Pharmacology, Study Chair — CMH Kharian Medical College
Locations (1):
- CMH Kharian Medical College, Kharan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided
The decision will be taken after getting consent from each participant.